CLINICAL TRIAL: NCT05567250
Title: Testing a Scalable Model For ACEs-Related Care Navigation Via 211 Telephone-Based Services
Brief Title: Testing a Scalable Model For ACEs-Related Care Navigation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Kaiser Permanente School of Medicine (Other)
Responsible Party: Principal Investigator, Rebecca Dudovitz, MD, MSHS, Associate Professor, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-000405
Record Dates: First submitted 2022-09-28; First posted 2022-10-05 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Adverse Childhood Experiences; Child Development
Keywords: Health Services Research; Care Coordination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Intervention + Usual Care (Experimental): Intervention group families will receive usual care and they will be connected via telephone to 211LA.
  Interventions: Behavioral: Behavioral: Telephone-based ACEs care coordination
- No Intervention: Usual Care (No Intervention): This group will receive usual care

INTERVENTIONS:
Behavioral: Behavioral: Telephone-based ACEs care coordination — The 211LA care coordinator will use the agency's extensive resource directory to identify and provide appropriate referral recommendations to each family. In addition, they will develop a care coordination plan, noting these recommendations and plans for follow-up, to be provided to the family's clinical care provider. The coordinator will routinely follow-up with the family until 1) children begin receiving services, 2) families refuse services, or 3) children are deemed ineligible by service providers.
  Arms: Experimental Intervention + Usual Care

SUMMARY:
The study is a randomized controlled trial of a telephone-based care coordination system for families who experienced Adverse Childhood Events (ACEs). The investigators will conduct the study in partnership with Kaiser Permanente School of Medicine (KPSOM) and 2-1-1 Los Angeles County (211LA), part of a national network of 2-1-1 call centers covering 93% of the US population. The study will test the effectiveness of 211LA in increasing referrals and services for families who screen positive for ACEs.

DETAILED DESCRIPTION:
The trial will enroll 200 children ages 0-11 years from the three FQHCs partner clinics, who screen positive for at least 1 ACE during their clinical encounter. The research study team will randomize children 1:1 into intervention (connection to 211LA for ACEs care coordination + usual care) or control (usual care alone).

Primary outcomes will include number of referrals to, eligibility for, and receipt of ACE-related services among intervention group participants compared to controls.

The investigators will measure these outcomes through parent reported data and 211LA data at baseline and 6 months after enrollment.

Expected findings include higher referral and service rates by six months after enrollment among intervention group participants.

ELIGIBILITY:
Inclusion Criteria:

* A patient in one of the three partner community clinic systems (ChapCare, Via Care and NEVHC)
* Child aged 0 - 11 years old
* Parent or legal guardian of child at least 18 years of age
* Comfortable completing a survey by interview in English or Spanish

Exclusion Criteria:

* Child or sibling already enrolled in this study
* Child or sibling enrolled in the AMP Child Development study

Max Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 102 (Actual)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-11-24 (Actual)

PRIMARY OUTCOMES:
Referrals to ACEs-related services | 2-6 months after enrollment
  The percentage of children who are referred to at least one ACEs-related service, as reported on the participant survey.

SECONDARY OUTCOMES:
Receipt of ACEs-related services | 2-6 months after enrollment
  The percentage of children who receive at least one ACEs-related service, as reported on the participant survey.
Number of referrals received | 2-6 months after enrollment
  The number of referrals made for ACEs-related services, as reported on the participant survey.
Number of services received | 2-6 months after enrollment
  The number of ACEs-related services received, as reported on the participant survey.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Dudovitz, MD MSHS, Principal Investigator — University of California, Los Angeles
Locations (1):
- University of California Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared within 2 years of study completion.
Access Criteria: Proposals should be directed to lporras@mednet.ucla.edu. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website, to be provided when requests are approved.

REFERENCES:
- [Background] Nelson BB, Thompson LR, Herrera P, Biely C, Arriola Zarate D, Aceves I, Estrada I, Chan V, Orantes C, Chung PJ. Telephone-Based Developmental Screening and Care Coordination Through 2-1-1: A Randomized Trial. Pediatrics. 2019 Apr;143(4):e20181064. doi: 10.1542/peds.2018-1064. PMID 30894408
- [Derived] Lim Chang C, Chung PJ, Ngan H, Porras-Javier L, Vangala S, Correa-Mendoza L, Calderon K, Thompson LR, Molina D, Aceves I, Torres F, Dudovitz R. Testing a Scalable Model for Adverse Childhood Experiences-Related Care Coordination via 211 Telephone-Based Services. Acad Pediatr. 2026 Jan-Feb;26(1):103160. doi: 10.1016/j.acap.2025.103160. Epub 2025 Oct 27. PMID 41161485